CLINICAL TRIAL: NCT07262593
Title: Family-Based Meal Timing for Cancer Prevention Among Native Hawaiian and Other Pacific Islanders: FAMTIME
Acronym: FAMTIME
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient metabolic kitchen support
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HCI166790
Record Dates: First submitted 2023-09-05; First posted 2025-12-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Cancer Prevention
Keywords: Diet; Time Restricted Eating; Quality of Life
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Participants received isocaloric, culturally tailored, pre-prepared meals to control underlying diet during TRE and control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Participants will continue their usual lifestyle.
- Time Restricted Eating (TRE) (Experimental): Participants will complete the TRE schedule for 8 weeks.
  Interventions: Other: Time Restricted Eating (TRE)
- Medically Tailored Meals (MTM) (Experimental): Participants will be given MTM for 8 weeks.
  Interventions: Other: Medically Tailored Meals (MTM)
- Time Restricted Eating (TRE) + Medically Tailored Meals (MTM) (Experimental): Participants will complete the TRE schedule and be given MTM for 8 weeks.
  Interventions: Other: Time Restricted Eating (TRE); Other: Medically Tailored Meals (MTM)

INTERVENTIONS:
Other: Time Restricted Eating (TRE) — For 8 weeks, participants will consume calorie containing foods and beverages within a personalized eating window up to 4-hours < baseline (e.g., 14-hr 10hr; 13hr 9-hr), but not >10-hours. Eating will start within 3-hours from waking and finish at least 3-hours before bedtime.
  Arms: Time Restricted Eating (TRE); Time Restricted Eating (TRE) + Medically Tailored Meals (MTM)
Other: Medically Tailored Meals (MTM) — For 8 weeks, participants will receive isocaloric, culturally tailored, nutritionally balanced lunch and dinner pre-prepared meals, plus a breakfast and snack menu that meets daily calorie requirements for weight maintenance.
  Arms: Medically Tailored Meals (MTM); Time Restricted Eating (TRE) + Medically Tailored Meals (MTM)

SUMMARY:
Native Hawaiian or other Pacific Islanders (NHPI) including those from Polynesia, Micronesia, and Melanesia, are the fastest growing racial/ethnic group in the U.S., but they are vastly underrepresented in health research. Compared with other racial/ethnic groups, NHPIs have higher risk of cancer, especially breast, colorectal and endometrial cancers. Moreover, NHPIs experience worse cancer-free survival, particularly among younger adults. There has been a concerning increase in incidence and deaths from cancer among NHPIs in recent years in parallel with persistent or widening health disparity gaps in cancer risk factors like poor diet quality, obesity, diabetes, and access to healthcare. Identifying culturally tailored ways to address these cancer risk factors in the NHPI community is therefore an urgent unmet need.

DETAILED DESCRIPTION:
Native Hawaiian and other Pacific Islanders (NHPI) from Polynesia, Micronesia, and Melanesia are the fastest growing racial/ethnic group in the U.S., but are vastly underrepresented in health research. NHPIs experience major disparities in risk of breast, colorectal, and endometrial cancers, and worse cancer-free survival, particularly among younger adults. There has been a concerning increase in cancer incidence and deaths among NHPIs in recent years in parallel with persistent or widening health disparity gaps in cancer risk factors like poor diet quality, obesity, diabetes, and access to healthcare. Identifying culturally tailored ways to address cancer risk factors in the NHPI community is therefore an urgent unmet need.

Diet is a cornerstone of managing metabolic health for cancer prevention. Irregular meal timing can disrupt 24-hour circadian clock-regulated metabolism to promote metabolic dysfunction, whereas structured mealtimes realign circadian transcriptional programs to improve metabolic health. Time restricted eating (TRE) is a form of intermittent fasting where daily calories are eaten within 6-12 hours. TRE improves cancer risk factors including hyperinsulinemia and dyslipidemia, but has not been evaluated in NHPIs. The investigators conducted a pilot 6-month randomized, controlled, crossover trial to test the feasibility and acceptability of TRE for effects on metabolic health in NHPIs at risk of endometrial cancer (TIMESPAN, NCT04763902). TIMESPAN was designed with feedback from focus groups and the Community Advisory Board (CAB) of NHPIs. Participants received isocaloric, culturally tailored, pre-prepared meals to control underlying diet during TRE and control. Insulin/c-peptide, triglycerides, and blood pressure improved with each phase, but TRE had larger effects and improved mood, energy, and satiety. The prepared meals addressed food insecurity and educated participants on healthy eating and portion control, goals of Medically Tailored Meals (MTM). A limitation was that the investigators did not measures effects of TRE without diet control. Since communal eating is integral to NHPI customs,13 participants reported that not providing family meals was a barrier.

The investigators propose to provide family meals and include a TRE arm without diet control in the, "Family-Based Meal Timing for Cancer Prevention among Native Hawaiian and other Pacific Islanders: FAMTIME" study. The long-term goal of this study is to address cancer risk disparities in NHPIs using diet strategies. The investigators will recruit 10 NHPI females at risk of obesity-related cancer (i.e., hyperglycemia, dyslipidemia, overweight/obese, history of diabetes, or cancer precursor lesions) who fast <12-hrs/day. Participants will complete a 2-week run-in period, then be randomized to 8-weeks' of (1) Control, (2) MTMs (healthy Polynesian diet), (3) TRE with usual diet, or (4) TRE + MTMs. Participants will also complete a 6-month follow-up. Family social support via communal eating will be encouraged. The myCircadianClock (mCC) app will evaluate and promote compliance. The central hypothesis is that MTM and TRE will improve metabolic and mental health among NHPI females at risk of obesity-related cancer; MTM+TRE will be multiplicative.

Aim 1. Determine the feasibility, fidelity and preliminary acceptability of TRE and MTM among Pacific Islander women at risk for developing endometrial cancer. Participants will be randomized using stratification by age group and BMI category to balance groups according to those variables. Feasibility will be evaluated by: (1) Proportion (%) of women referred that were recruited and consented; (2) attrition as a function of time; (3) % of scheduled biospecimen collections and questionnaires completed; (4) number of TRE or MTM adherent days per week (participants will be considered adherent if they fasted between 14-18 h per day during the TRE phase according to mealtime log); (5) % meals delivered on schedule. The study will be considered feasible if >70% women are consented and retained, complete all biospecimen collections and questionnaires, and if women adhere to the TRE protocol for at least 5/7 days per week. Fidelity will be evaluated as % protocol checklist items delivered as intended with a goal of 90%.

Aim 2. Compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer. Primary outcome: hyperinsulinemia (C-peptide). Secondary outcomes: waist/hip ratio, weight, body composition, c-reactive protein, fasting glucose/insulin, 24-hour glucose, HOMA-IR, atherogenic lipids, blood pressure, blood metabolites related to cancer risk, appetite, diet quality, sleep quality/duration, and physical activity.

Aim 3. Compare TRE, MTM, TRE + MTM, and Control for effects on emotional wellbeing among NHPI women at risk of obesity-related cancer. Focus groups and the CAB reported that mental wellbeing is the most important outcome to NHPI women, yet it is rarely discussed or evaluated. The primary outcome is depression (PHQ-9). Secondary outcomes: anxiety, alcohol use, health status, social support, and acculturative stress. These outcome measures were endorsed by the CAB as being particularly relevant.

Aim 4. Qualitatively investigate the roles of social support and mental health in diet behavior change among NHPI women at risk of obesity-related cancer and their household. The investigators will build upon the themes that emerged from TIMESPAN by conducting focus groups among (1) FAMTIME participants and their household members, (2) the CAB, to interpret outcomes and evaluate the intervention from a cultural perspective. The investigators will explore in-depth the roles of social support, mental health, and food security in behavior change, and how to optimize cancer prevention interventions for high impact in the NHPI community.

ELIGIBILITY:
Inclusion Criteria:

1. Native Hawaiian/Pacific Islander females aged 18 years or older
2. Have at least one cancer risk factor (BMI≥25kg/m2 OR have a history of non-insulin dependent diabetes OR have at least one metabolic syndrome criteria out of clinical range OR have a history of cancer precursors (e.g., atypical endometrial hyperplasia, colorectal adenoma, atypical ductal hyperplasia)
3. Have a working cell phone that can download an App
4. Able to use cell phone during day (e.g. at work)
5. Not a night shift worker
6. Able to attend study visits at the Huntsman Cancer Institute Center for HOPE
7. Not on a special diet
8. Fast <14-hours per night (i.e., eat all calorie containing foods over >10-hours/day)

Exclusion Criteria:

1. Unable to provide informed consent
2. Necessity of a special diet
3. Have a history of insulin dependent diabetes
4. Have a history of hysterectomy
5. Fast >14-hours per night/<10-hour eating window

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Proportion of women recruited/consented - Feasibility | From enrollment to the 6-month follow up survey.
  To determine the feasibility, fidelity, and preliminary acceptability of TRE and MTM among Pacific Islander women at risk for developing endometrial cancer.
  This outcome measure will report the proportion of women referred who were recruited and consented to the trial. The study will be considered feasible if >70% of women approached consent to the study.
C-Peptide - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  Hyperinsulinemia is a condition of too much insulin in the blood and is a cancer risk factor. C-peptide measures the amount of C-peptide in the blood and is an indicator of hyperinsulinemia.
  This outcome measure will report the mean C-peptide of each group at 8 weeks after the initiation of the intervention.
Depression - Emotional well-being | From enrollment to the 6 month follow up survey
  To compare TRE, MTM, TRE + MTM, and Control for effects on emotional well-being among NHPI women at risk of obesity-related cancer.
  Depression will be assessed with the Patient Health Questionnaire (PHQ-9). Scores range from 1-27, with lower scores indicating minimal depression and higher scores indicating more severe depression. A reduction of 5 points is considered clinically meaningful. This outcome measure will report the mean PHQ-9 scale of each group at 8 weeks after the initiation of the intervention.

SECONDARY OUTCOMES:
Attrition - Feasibility | From enrollment to the 6 month follow up survey
  To determine the feasibility, fidelity, and preliminary acceptability of TRE and MTM among Pacific Islander women at risk for developing endometrial cancer.
  This outcome measure will report the study's attrition, or the number of participants who drop out of this trial after randomization. The study will be considered feasible if >70% of women randomized complete the study.
Study Procedures Completed - Feasibility | From enrollment to the 6 month follow up survey
  To determine the feasibility, fidelity, and preliminary acceptability of TRE and MTM among Pacific Islander women at risk for developing endometrial cancer.
  This outcome measure will report the proportion of scheduled biospecimen collections and questionnaires that were completed. The study will be considered feasible if study participants complete 100% of biospecimen collections and questionnaires.
TRE Adherent Days - Feasibility | From enrollment to the 6 month follow up survey
  To determine the feasibility, fidelity, and preliminary acceptability of TRE and MTM among Pacific Islander women at risk for developing endometrial cancer.
  This outcome measure will report the mean number of TRE or MTM adherent days per week. Participants will be considered adherent if they fasted between 14-18 h per day during the TRE phase according to mealtime log. The study will be considered feasible if participants adhere to the TRE protocol for at least 5/7 days per week.
Meals Delivered - Feasibility | From enrollment to the 6 month follow up survey
  To determine the feasibility, fidelity, and preliminary acceptability of TRE and MTM among Pacific Islander women at risk for developing endometrial cancer.
  This outcome measure will report the proportion of meals delivered on schedule. Fidelity will be evaluated as % protocol checklist items delivered as intended with a goal of 90%.
Protocol Items Delivered as Intended - Fidelity | From enrollment to the 6 month follow up survey
  To determine the feasibility, fidelity, and preliminary acceptability of TRE and MTM among Pacific Islander women at risk for developing endometrial cancer.
  This outcome measure will report the proportion of protocol checklist items delivered as intended. Fidelity will be achieved if 90% of protocol checklist items are delivered as intended.
Waist/hip - Effects on Metabolic Cancer Risk | From enrollment to the 6 month follow up survey
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  Waist/hip ratio is waist circumference divided by hip circumference. This outcome measure will report the mean waist/hip ratio of each group at 8 weeks after the initiation of the intervention.
Weight - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  This outcome measure will report the mean weight ratio of each group at 8 weeks after the initiation of the intervention.
Body composition - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  Body composition is the percentage (%) of weight that is fat tissue. This outcome measure will report the mean body composition of each group at 8 weeks after the initiation of the intervention.
C-reactive protein - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  C-reactive protein (CRP) is the amount of a protein made by the liver. CRP is a risk of obesity-related cancer. This outcome measure will report the mean CRP of each group at 8 weeks after the initiation of the intervention.
Fasting glucose - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  Fasting glucose is the amount of glucose in the blood after abstaining from food for 8 hours. This outcome measure will report the mean fasting glucose of each group at 8 weeks after the initiation of the intervention.
Fasting insulin - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  Fasting glucose is the amount of insulin in the blood after abstaining from food for 8 hours. This outcome measure will report the mean fasting insulin of each group at 8 weeks after the initiation of the intervention.
24-hour glucose - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  24-hour glucose is the mean glucose in the blood over 24 hours. This outcome measure will report the mean 24-hour glucose of each group at 8 weeks after the initiation of the intervention.
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  HOMA-IR is an equation used to quantify insulin resistance. This outcome measure will report the mean HOMA-IR of each group at 8 weeks after the initiation of the intervention.
Low-density lipoprotein (LDL) - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  Low-density lipoprotein (LDL) is an atherogenic lipid that is a risk of obesity-related cancer. This outcome measure will report the mean LDL of each group at 8 weeks after the initiation of the intervention.
Blood pressure - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  This outcome measure will report the mean blood pressure of each group at 8 weeks after the initiation of the intervention.
Lipidomics - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  This outcome measure will report the lipidomics of each group at 8 weeks after the initiation of the intervention.
Metabolomics - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  This outcome measure will report the metabolomics of each group at 8 weeks after the initiation of the intervention.
Appetite - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  Appetite will be measured as a single self-reported item. This outcome measure will report the responses of each group at 8 weeks after the initiation of the intervention.
Diet quality - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  Diet quality will be assess by the Healthy Eating Index (HEI)-2020 and assessed via 24-hour recall.
  The HEI-2020 score is a quantification of well diet aligns with the Dietary Guidelines for Americans. HEI-2020 has a maximum total score of 100 and a minimum score of 0, with higher scores indicating better alignment with dietary guidelines and lower scores indicating poorer alignment.
  This outcome measure will report the mean HEI-2020 of each group at 8 weeks after the initiation of the intervention.
Sleep Quality - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  Sleep quality will be measured as a single, self-reported item on a survey. This outcome measure will report the count of responses from each group at 6 months after the initiation of the intervention.
Sleep Duration - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  Sleep duration will be objectively measured on a research-grade accelerometer worn on the wrist. This outcome measure will report the mean sleep duration of each group at 8 weeks after the initiation of the intervention.
Physical Activity - Effects on Metabolic Cancer Risk | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on metabolic cancer risk factors among NHPI women at risk of obesity-related cancer.
  Physical activity will be objectively measured on a research-grade accelerometer worn on the wrist. This outcome measure will report the mean daily steps of each group at 8 weeks after the initiation of the intervention.
Anxiety - Emotional Well-being | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on emotional well-being among NHPI women at risk of obesity-related cancer.
  Anxiety will be assessed with the Generalized Anxiety Disorder 7-item survey (GAD-7). Scores range from 0-15, with lower scores indicating minimal anxiety and higher scores indicating more severe anxiety.
  This outcome measure will report the mean GAD-7 score of each group at 8 weeks after the initiation of the intervention.
Alcohol Use - Emotional Well-being | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on emotional well-being among NHPI women at risk of obesity-related cancer.
  Alcohol use will be assessed with the Alcohol use disorders identification test (AUDIT-C). Scores range from 0-12, with lower scores indicating minimal alcohol use and higher scores indicating more severe alcohol use.
  This outcome measure will report the mean AUDIT-C score of each group at 8 weeks after the initiation of the intervention.
Health status - Emotional Well-being | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on emotional well-being among NHPI women at risk of obesity-related cancer.
  Health status will be assessed by a single, self-reported item. Subject will be asked to report their general health status from 1, Excellent to 5, Poor
  This outcome measure will report the count of participants selecting each response at 6 months after the initiation of the intervention.
Acculturative stress - Emotional Well-being | From enrollment to the 6-month follow up survey.
  To compare TRE, MTM, TRE + MTM, and Control for effects on emotional well-being among NHPI women at risk of obesity-related cancer.
  Acculturative stress will be assessed with the Pacific Islands cultural orientation acculturative stress survey (PIACCULT). This is a self reported, 11-item assessment.
  Scores range from 11-55, with lower scores indicating worse Pacific cultural orientation and higher scores indicating more Pacific cultural orientation.
  This outcome measure will report the mean PIACCULT score of each group at 6 months after the initiation of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Playdon, PhD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ethoan LN, Takata Y, Sakuma KK, Irvin VL. Trends in Clinical Research Including Asian American, Native Hawaiian, and Pacific Islander Participants Funded by the US National Institutes of Health, 1992 to 2018. JAMA Netw Open. 2019 Jul 3;2(7):e197432. doi: 10.1001/jamanetworkopen.2019.7432. PMID 31339543
- [Background] Liu L, Noone AM, Gomez SL, Scoppa S, Gibson JT, Lichtensztajn D, Fish K, Wilkens LR, Goodman MT, Morris C, Kwong S, Deapen D, Miller BA. Cancer incidence trends among native Hawaiians and other Pacific Islanders in the United States, 1990-2008. J Natl Cancer Inst. 2013 Aug 7;105(15):1086-95. doi: 10.1093/jnci/djt156. Epub 2013 Jul 22. PMID 23878354
- [Background] Terada K, Carney M, Kim R, Ahn HJ, Miyamura J. Health Disparities in Native Hawaiians and Other Pacific Islanders Following Hysterectomy for Endometrial Cancer. Hawaii J Med Public Health. 2016 May;75(5):137-9. PMID 27239393
- [Background] Kost ER, Hall KL, Hines JF, Farley JH, Nycum LR, Rose GS, Carlson JW, Fischer JR Jr, Kendall BS. Asian-Pacific Islander race independently predicts poor outcome in patients with endometrial cancer. Gynecol Oncol. 2003 May;89(2):218-26. doi: 10.1016/s0090-8258(03)00050-7. PMID 12713983
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Equity. OoH. Twenty years of health data for Native Hawaiian/Pacific Islander communities in Utah. Salt Lake City, UT: 2023.
- [Background] Subica AM, Agarwal N, Sullivan JG, Link BG. Obesity and Associated Health Disparities Among Understudied Multiracial, Pacific Islander, and American Indian Adults. Obesity (Silver Spring). 2017 Dec;25(12):2128-2136. doi: 10.1002/oby.21954. Epub 2017 Oct 25. PMID 29071803
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in body-mass index, underweight, overweight, and obesity from 1975 to 2016: a pooled analysis of 2416 population-based measurement studies in 128.9 million children, adolescents, and adults. Lancet. 2017 Dec 16;390(10113):2627-2642. doi: 10.1016/S0140-6736(17)32129-3. Epub 2017 Oct 10. PMID 29029897
- [Background] Research. WCRFAIfC. Continuous Update Project Expert Report 2018 2018 [Accessed 10th September, 2023]. Available from: Available at dietandcancerreport.org
- [Background] Petersen MC, Gallop MR, Flores Ramos S, Zarrinpar A, Broussard JL, Chondronikola M, Chaix A, Klein S. Complex physiology and clinical implications of time-restricted eating. Physiol Rev. 2022 Oct 1;102(4):1991-2034. doi: 10.1152/physrev.00006.2022. Epub 2022 Jul 14. PMID 35834774
- [Background] Chaix A, Manoogian ENC, Melkani GC, Panda S. Time-Restricted Eating to Prevent and Manage Chronic Metabolic Diseases. Annu Rev Nutr. 2019 Aug 21;39:291-315. doi: 10.1146/annurev-nutr-082018-124320. Epub 2019 Jun 10. PMID 31180809
- [Background] Downer S, Berkowitz SA, Harlan TS, Olstad DL, Mozaffarian D. Food is medicine: actions to integrate food and nutrition into healthcare. BMJ. 2020 Jun 29;369:m2482. doi: 10.1136/bmj.m2482. PMID 32601089
- [Background] Playdon M, Rogers TN, Brooks E, Petersen EM, Tavake-Pasi F, Lopez JA, Quintana X, Aitaoto N, Rogers CR. Sociocultural influences on dietary behavior and meal timing among Native Hawaiian and Pacific Islander women at risk of endometrial cancer: a qualitative investigation. Cancer Causes Control. 2023 Jan;34(1):23-37. doi: 10.1007/s10552-022-01628-0. Epub 2022 Oct 8. PMID 36208351
- [Background] Bidonde J, Fagerlund BC, Fronsdal KB, Lund UH, Robberstad B. FreeStyle Libre Flash Glucose Self-Monitoring System: A Single-Technology Assessment [Internet]. Oslo, Norway: Knowledge Centre for the Health Services at The Norwegian Institute of Public Health (NIPH); 2017 Aug 21. Report from the Norwegian Institute of Public Health No. 2017-07. Available from http://www.ncbi.nlm.nih.gov/books/NBK482068/ PMID 29553668
- [Background] Muniyappa R, Madan R, Varghese RT. Assessing Insulin Sensitivity and Resistance in Humans. 2024 Oct 16. In: Feingold KR, Adler RA, Ahmed SF, Anawalt B, Blackman MR, Chrousos G, Corpas E, de Herder WW, Dhatariya K, Dungan K, Hamilton E, Hofland J, Jan de Beur S, Kalra S, Kaltsas G, Kapoor N, Kim M, Koch C, Kopp P, Korbonits M, Kovacs CS, Kuohung W, Laferrere B, Levy M, McGee EA, McLachlan R, Muzumdar R, Purnell J, Rey R, Sahay R, Shah AS, Sperling MA, Stratakis CA, Trence DL, Wilson DP, editors. Endotext [Internet]. South Dartmouth (MA): MDText.com, Inc.; 2000-. Available from http://www.ncbi.nlm.nih.gov/books/NBK278954/ PMID 25905189
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749
- [Background] Shams-White MM, Pannucci TE, Lerman JL, Herrick KA, Zimmer M, Meyers Mathieu K, Stoody EE, Reedy J. Healthy Eating Index-2020: Review and Update Process to Reflect the Dietary Guidelines for Americans,2020-2025. J Acad Nutr Diet. 2023 Sep;123(9):1280-1288. doi: 10.1016/j.jand.2023.05.015. Epub 2023 May 16. PMID 37201748
- [Background] Subar AF, Kirkpatrick SI, Mittl B, Zimmerman TP, Thompson FE, Bingley C, Willis G, Islam NG, Baranowski T, McNutt S, Potischman N. The Automated Self-Administered 24-hour dietary recall (ASA24): a resource for researchers, clinicians, and educators from the National Cancer Institute. J Acad Nutr Diet. 2012 Aug;112(8):1134-7. doi: 10.1016/j.jand.2012.04.016. Epub 2012 Jun 15. No abstract available. PMID 22704899
- [Background] Keadle SK, Patel S, Berrigan D, Christopher CN, Huang J, Saint-Maurice PF, Loftfield E, Matthews CE. Validation of ACT24 Version 2.0 for Estimating Behavioral Domains, Active and Sedentary Time. Med Sci Sports Exerc. 2023 Jun 1;55(6):1054-1062. doi: 10.1249/MSS.0000000000003135. Epub 2023 Jan 29. PMID 36719650
- [Background] Activinsights. GENEActiv: Raw Data Accelerometry 2023 [cited Accessed 16th September, 2023]. Available from: https://activinsights.com/technology/geneactiv/.
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Subica AM, Aitaoto N, Link BG, Yamada AM, Henwood BF, Sullivan G. Mental Health Status, Need, and Unmet Need for Mental Health Services Among U.S. Pacific Islanders. Psychiatr Serv. 2019 Jul 1;70(7):578-585. doi: 10.1176/appi.ps.201800455. Epub 2019 Apr 17. PMID 30991907
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Bush K, Kivlahan DR, McDonell MB, Fihn SD, Bradley KA. The AUDIT alcohol consumption questions (AUDIT-C): an effective brief screening test for problem drinking. Ambulatory Care Quality Improvement Project (ACQUIP). Alcohol Use Disorders Identification Test. Arch Intern Med. 1998 Sep 14;158(16):1789-95. doi: 10.1001/archinte.158.16.1789. PMID 9738608
- [Background] (CDC). CfDCaP. Behavioral Risk Factor Surveillance System Survey Questionnaire tlanta, Georgia2022 [Accessed 10th September, 2023]. Available from: https://www.cdc.gov/brfss/questionnaires/index.htm.
- [Background] Manuela S, Sibley CG. The Pacific Identity and Wellbeing Scale-Revised (PIWBS-R). Cultur Divers Ethnic Minor Psychol. 2015 Jan;21(1):146-55. doi: 10.1037/a0037536. Epub 2014 Aug 11. PMID 25111555
- [Background] Schluter PJ, Tautolo el-S, Paterson J. Acculturation of Pacific mothers in New Zealand over time: findings from the Pacific Islands Families study. BMC Public Health. 2011 May 12;11:307. doi: 10.1186/1471-2458-11-307. PMID 21569444
- [Background] Nguyen-Truong CKY, Waters SF, Richardson M, Barrow N, Seia J, Eti DU, Rodela KF. An Antiracism Community-Based Participatory Research With Organizations Serving Immigrant and Marginalized Communities, Including Asian Americans and Native Hawaiians/Pacific Islanders in the United States Pacific Northwest: Qualitative Description Study With Key Informants. Asian Pac Isl Nurs J. 2023 Jan 11;7:e43150. doi: 10.2196/43150. PMID 36648292
- [Background] Taparra K, Harding M, Deville C. Healing and Health Equity for Asian American, Native Hawaiian, and Pacific Islander Populations. JAMA. 2021 Dec 21;326(23):2432-2433. doi: 10.1001/jama.2021.19243. No abstract available. PMID 34932087
- [Background] Office of Health Disparities. Utah Health Status by Race and Ethnicity 2021. Salt Lake City, UT: Utah Department of Health.
- [Background] Moy KL, Sallis JF, David KJ. Health indicators of Native Hawaiian and Pacific Islanders in the United States. J Community Health. 2010 Feb;35(1):81-92. doi: 10.1007/s10900-009-9194-0. PMID 19856087
- [Background] Harry ML, Sanchez K, Ahmedani BK, Beck AL, Coleman KJ, Coley RY, Daida YG, Lynch FL, Rossom RC, Waring SC, Simon GE. Assessing the differential item functioning of PHQ-9 items for diverse racial and ethnic adults with mental health and/or substance use disorder diagnoses: A retrospective cohort study. J Affect Disord. 2023 Oct 1;338:402-413. doi: 10.1016/j.jad.2023.04.091. Epub 2023 Apr 29. PMID 37127116
- [Background] Hooker K, Phibbs S, Irvin VL, Mendez-Luck CA, Doan LN, Li T, Turner S, Choun S. Depression Among Older Adults in the United States by Disaggregated Race and Ethnicity. Gerontologist. 2019 Sep 17;59(5):886-891. doi: 10.1093/geront/gny159. PMID 30561600
- [Background] Alhomsi A, Strassle PD, Ponce S, Mendez I, Quintero SM, Wilkerson M, Stewart AL, Napoles AM. Financial Hardship and Psychological Distress During the Pandemic: A Nationally Representative Survey of Major Racial-Ethnic Groups in the United States. Health Equity. 2023 Jul 20;7(1):395-405. doi: 10.1089/heq.2022.0197. eCollection 2023. PMID 37483650
- [Background] Kwan PP, Pike JR, Co DE, Esmundo S, Vaivao DES, May VT, Pang JK, Sabado-Liwag M, Tan NS, Tanjasiri SP, Xie B, Palmer PH. Association Between Stress and Social Support Among Young Adult Pacific Islander Smokers. Hawaii J Health Soc Welf. 2023 Feb;82(2):31-38. PMID 36779006
- [Background] McLaughlin LA, Braun KL. Asian and Pacific Islander cultural values: considerations for health care decision making. Health Soc Work. 1998 May;23(2):116-26. doi: 10.1093/hsw/23.2.116. PMID 9598394
- [Background] Subica AM, Aitaoto N, Sullivan JG, Henwood BF, Yamada AM, Link BG. Mental illness stigma among Pacific Islanders. Psychiatry Res. 2019 Mar;273:578-585. doi: 10.1016/j.psychres.2019.01.077. Epub 2019 Jan 26. PMID 30716597
- [Background] Clarke MA, Devesa SS, Harvey SV, Wentzensen N. Hysterectomy-Corrected Uterine Corpus Cancer Incidence Trends and Differences in Relative Survival Reveal Racial Disparities and Rising Rates of Nonendometrioid Cancers. J Clin Oncol. 2019 Aug 1;37(22):1895-1908. doi: 10.1200/JCO.19.00151. Epub 2019 May 22. PMID 31116674
- [Background] Sheikh MA, Althouse AD, Freese KE, Soisson S, Edwards RP, Welburn S, Sukumvanich P, Comerci J, Kelley J, LaPorte RE, Linkov F. USA endometrial cancer projections to 2030: should we be concerned? Future Oncol. 2014 Dec;10(16):2561-8. doi: 10.2217/fon.14.192. PMID 25531045
- [Background] Ferlay J, Steliarova-Foucher E, Lortet-Tieulent J, Rosso S, Coebergh JW, Comber H, Forman D, Bray F. Cancer incidence and mortality patterns in Europe: estimates for 40 countries in 2012. Eur J Cancer. 2013 Apr;49(6):1374-403. doi: 10.1016/j.ejca.2012.12.027. Epub 2013 Feb 26. PMID 23485231
- [Background] Esposito K, Chiodini P, Colao A, Lenzi A, Giugliano D. Metabolic syndrome and risk of cancer: a systematic review and meta-analysis. Diabetes Care. 2012 Nov;35(11):2402-11. doi: 10.2337/dc12-0336. PMID 23093685
- [Background] Esposito K, Chiodini P, Capuano A, Bellastella G, Maiorino MI, Giugliano D. Metabolic syndrome and endometrial cancer: a meta-analysis. Endocrine. 2014 Feb;45(1):28-36. doi: 10.1007/s12020-013-9973-3. Epub 2013 May 3. PMID 23640372
- [Background] World Cancer Research Fund/American Institute for Cancer Research. Diet, Nutrition, Physical Activity and Cancer: a Global Perspective. Continuous Update Project Report 2018. 2018.
- [Background] Michels KA, McNeel TS, Trabert B. Metabolic syndrome and risk of ovarian and fallopian tube cancer in the United States: An analysis of linked SEER-Medicare data. Gynecol Oncol. 2019 Nov;155(2):294-300. doi: 10.1016/j.ygyno.2019.08.032. Epub 2019 Sep 5. PMID 31495456
- [Background] Karra P, Winn M, Pauleck S, Bulsiewicz-Jacobsen A, Peterson L, Coletta A, Doherty J, Ulrich CM, Summers SA, Gunter M, Hardikar S, Playdon MC. Metabolic dysfunction and obesity-related cancer: Beyond obesity and metabolic syndrome. Obesity (Silver Spring). 2022 Jul;30(7):1323-1334. doi: 10.1002/oby.23444. PMID 35785479
- [Background] Stocks T, Bjorge T, Ulmer H, Manjer J, Haggstrom C, Nagel G, Engeland A, Johansen D, Hallmans G, Selmer R, Concin H, Tretli S, Jonsson H, Stattin P. Metabolic risk score and cancer risk: pooled analysis of seven cohorts. Int J Epidemiol. 2015 Aug;44(4):1353-63. doi: 10.1093/ije/dyv001. Epub 2015 Feb 3. PMID 25652574
- [Background] Ahern TP, Hankinson SE, Willett WC, Pollak MN, Eliassen AH, Tamimi RM. Plasma C-peptide, mammographic breast density, and risk of invasive breast cancer. Cancer Epidemiol Biomarkers Prev. 2013 Oct;22(10):1786-96. doi: 10.1158/1055-9965.EPI-13-0375. PMID 24097198
- [Background] Kliemann N, Ould Ammar R, Biessy C, Gicquiau A, Katzke V, Kaaks R, Tjonneland A, Olsen A, Sanchez MJ, Crous-Bou M, Pasanisi F, Tin Tin S, Perez-Cornago A, Aune D, Christakoudi S, Heath AK, Colorado-Yohar SM, Grioni S, Skeie G, Sartor H, Idahl A, Rylander C, May AM, Weiderpass E, Freisling H, Playdon MC, Rinaldi S, Murphy N, Huybrechts I, Dossus L, Gunter MJ. Metabolically Defined Body Size Phenotypes and Risk of Endometrial Cancer in the European Prospective Investigation into Cancer and Nutrition (EPIC). Cancer Epidemiol Biomarkers Prev. 2022 Jul 1;31(7):1359-1367. doi: 10.1158/1055-9965.EPI-22-0160. PMID 35437568
- [Background] Hernandez AV, Pasupuleti V, Benites-Zapata VA, Thota P, Deshpande A, Perez-Lopez FR. Insulin resistance and endometrial cancer risk: A systematic review and meta-analysis. Eur J Cancer. 2015 Dec;51(18):2747-58. doi: 10.1016/j.ejca.2015.08.031. Epub 2015 Nov 18. PMID 26597445
- [Background] Kitson SJ, Evans DG, Crosbie EJ. Identifying High-Risk Women for Endometrial Cancer Prevention Strategies: Proposal of an Endometrial Cancer Risk Prediction Model. Cancer Prev Res (Phila). 2017 Jan;10(1):1-13. doi: 10.1158/1940-6207.CAPR-16-0224. Epub 2016 Dec 13. PMID 27965288
- [Background] Shen J, Hernandez D, Ye Y, Wu X, Chow WH, Zhao H. Metabolic hormones and breast cancer risk among Mexican American Women in the Mano a Mano Cohort Study. Sci Rep. 2019 Jul 10;9(1):9989. doi: 10.1038/s41598-019-46429-9. PMID 31292496
- [Background] Wang Q, Tu H, Zhu M, Liang D, Ye Y, Chang DW, Long Y, Wu X. Circulating obesity-driven biomarkers are associated with risk of clear cell renal cell carcinoma: a two-stage, case-control study. Carcinogenesis. 2019 Oct 16;40(10):1191-1197. doi: 10.1093/carcin/bgz074. PMID 31001636
- [Background] Hidaka A, Budhathoki S, Yamaji T, Sawada N, Tanaka-Mizuno S, Kuchiba A, Charvat H, Goto A, Shimazu T, Inoue M, Noda M, Tsugane S, Iwasaki M; JPHC Study Group. Plasma C-peptide and glycated albumin and subsequent risk of cancer: From a large prospective case-cohort study in Japan. Int J Cancer. 2019 Feb 15;144(4):718-729. doi: 10.1002/ijc.31847. Epub 2018 Oct 30. PMID 30183080
- [Background] Liao LM, Hofmann JN, Cho E, Pollak MN, Chow WH, Purdue MP. Circulating levels of obesity-related markers and risk of renal cell carcinoma in the PLCO cancer screening trial. Cancer Causes Control. 2017 Jul;28(7):801-807. doi: 10.1007/s10552-017-0901-3. Epub 2017 May 8. PMID 28484923
- [Background] Gaudet MM, Patel AV, Teras LR, Sun J, Campbell PT, Stevens VL, Jacobs EJ, Gapstur SM. Obesity-related markers and breast cancer in CPS-II Nutrition Cohort. Int J Mol Epidemiol Genet. 2013 Sep 12;4(3):156-66. eCollection 2013. PMID 24046808
- [Background] Dallal CM, Brinton LA, Bauer DC, Buist DS, Cauley JA, Hue TF, Lacroix A, Tice JA, Chia VM, Falk R, Pfeiffer R, Pollak M, Veenstra TD, Xu X, Lacey JV Jr; B~FIT Research Group. Obesity-related hormones and endometrial cancer among postmenopausal women: a nested case-control study within the B~FIT cohort. Endocr Relat Cancer. 2013 Feb 18;20(1):151-60. doi: 10.1530/ERC-12-0229. Print 2013 Feb. PMID 23222000
- [Background] Jones AG, Hattersley AT. The clinical utility of C-peptide measurement in the care of patients with diabetes. Diabet Med. 2013 Jul;30(7):803-17. doi: 10.1111/dme.12159. PMID 23413806
- [Background] Babio N, Toledo E, Estruch R, Ros E, Martinez-Gonzalez MA, Castaner O, Bullo M, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Sorli JV, Salas-Salvado J; PREDIMED Study Investigators. Mediterranean diets and metabolic syndrome status in the PREDIMED randomized trial. CMAJ. 2014 Nov 18;186(17):E649-57. doi: 10.1503/cmaj.140764. Epub 2014 Oct 14. PMID 25316904
- [Background] World Cancer Research Fund International/American Institute for Cancer Research. World Cancer Research Fund International/American Institute for Cancer Research Continuous Update Project Report: Diet, Nutrition, Physical Activity, and Breast Cancer Survivors. 2014.
- [Background] Lemstra M, Bird Y, Nwankwo C, Rogers M, Moraros J. Weight loss intervention adherence and factors promoting adherence: a meta-analysis. Patient Prefer Adherence. 2016 Aug 12;10:1547-59. doi: 10.2147/PPA.S103649. eCollection 2016. PMID 27574404
- [Background] Dombrowski SU, Knittle K, Avenell A, Araujo-Soares V, Sniehotta FF. Long term maintenance of weight loss with non-surgical interventions in obese adults: systematic review and meta-analyses of randomised controlled trials. BMJ. 2014 May 14;348:g2646. doi: 10.1136/bmj.g2646. PMID 25134100
- [Background] Loveman E, Frampton GK, Shepherd J, Picot J, Cooper K, Bryant J, Welch K, Clegg A. The clinical effectiveness and cost-effectiveness of long-term weight management schemes for adults: a systematic review. Health Technol Assess. 2011 Jan;15(2):1-182. doi: 10.3310/hta15020. PMID 21247515
- [Background] Varkevisser RDM, van Stralen MM, Kroeze W, Ket JCF, Steenhuis IHM. Determinants of weight loss maintenance: a systematic review. Obes Rev. 2019 Feb;20(2):171-211. doi: 10.1111/obr.12772. Epub 2018 Oct 16. PMID 30324651
- [Background] O'Connor SG, Boyd P, Bailey CP, Shams-White MM, Agurs-Collins T, Hall K, Reedy J, Sauter ER, Czajkowski SM. Perspective: Time-Restricted Eating Compared with Caloric Restriction: Potential Facilitators and Barriers of Long-Term Weight Loss Maintenance. Adv Nutr. 2021 Mar 31;12(2):325-333. doi: 10.1093/advances/nmaa168. PMID 33463673
- [Background] Chlebowski RT, Reeves MM. Weight Loss Randomized Intervention Trials in Female Cancer Survivors. J Clin Oncol. 2016 Dec 10;34(35):4238-4248. doi: 10.1200/JCO.2016.69.4026. Epub 2016 Nov 7. PMID 27903147
- [Background] Aitaoto N, Campo S, Snetselaar LG, Janz KF, Farris KB, Parker E, Belyeu-Camacho T, Jimenez RP. Formative Research to Inform Nutrition Interventions in Chuuk and the US Pacific. J Acad Nutr Diet. 2015 Jun;115(6):947-53. doi: 10.1016/j.jand.2014.11.018. Epub 2015 Jan 27. PMID 25634092
- [Background] Stevens RG, Hansen J, Costa G, Haus E, Kauppinen T, Aronson KJ, Castano-Vinyals G, Davis S, Frings-Dresen MH, Fritschi L, Kogevinas M, Kogi K, Lie JA, Lowden A, Peplonska B, Pesch B, Pukkala E, Schernhammer E, Travis RC, Vermeulen R, Zheng T, Cogliano V, Straif K. Considerations of circadian impact for defining 'shift work' in cancer studies: IARC Working Group Report. Occup Environ Med. 2011 Feb;68(2):154-62. doi: 10.1136/oem.2009.053512. Epub 2010 Oct 20. PMID 20962033
- [Background] Gu F, Xu S, Devesa SS, Zhang F, Klerman EB, Graubard BI, Caporaso NE. Longitude Position in a Time Zone and Cancer Risk in the United States. Cancer Epidemiol Biomarkers Prev. 2017 Aug;26(8):1306-1311. doi: 10.1158/1055-9965.EPI-16-1029. Epub 2017 Apr 27. PMID 28450580
- [Background] Savvidis C, Koutsilieris M. Circadian rhythm disruption in cancer biology. Mol Med. 2012 Dec 6;18(1):1249-60. doi: 10.2119/molmed.2012.00077. PMID 22811066
- [Background] Shih MC, Yeh KT, Tang KP, Chen JC, Chang JG. Promoter methylation in circadian genes of endometrial cancers detected by methylation-specific PCR. Mol Carcinog. 2006 Oct;45(10):732-40. doi: 10.1002/mc.20198. PMID 16683245
- [Background] Patterson RE, Laughlin GA, LaCroix AZ, Hartman SJ, Natarajan L, Senger CM, Martinez ME, Villasenor A, Sears DD, Marinac CR, Gallo LC. Intermittent Fasting and Human Metabolic Health. J Acad Nutr Diet. 2015 Aug;115(8):1203-12. doi: 10.1016/j.jand.2015.02.018. Epub 2015 Apr 6. No abstract available. PMID 25857868
- [Background] Almoosawi S, Vingeliene S, Gachon F, Voortman T, Palla L, Johnston JD, Van Dam RM, Darimont C, Karagounis LG. Chronotype: Implications for Epidemiologic Studies on Chrono-Nutrition and Cardiometabolic Health. Adv Nutr. 2019 Jan 1;10(1):30-42. doi: 10.1093/advances/nmy070. PMID 30500869
- [Background] Codoner-Franch P, Gombert M, Martinez-Raga J, Cenit MC. Circadian Disruption and Mental Health: The Chronotherapeutic Potential of Microbiome-Based and Dietary Strategies. Int J Mol Sci. 2023 Apr 20;24(8):7579. doi: 10.3390/ijms24087579. PMID 37108739
- [Background] Luo J, Hendryx M, Manson JE, Figueiredo JC, LeBlanc ES, Barrington W, Rohan TE, Howard BV, Reding K, Ho GY, Garcia DO, Chlebowski RT. Intentional Weight Loss and Obesity-Related Cancer Risk. JNCI Cancer Spectr. 2019 Aug 9;3(4):pkz054. doi: 10.1093/jncics/pkz054. eCollection 2019 Dec. PMID 31737862
- [Background] Pan K, Luo J, Aragaki AK, Chlebowski RT. Weight loss, diet composition and breast cancer incidence and outcome in postmenopausal women. Oncotarget. 2019 May 3;10(33):3088-3092. doi: 10.18632/oncotarget.26864. eCollection 2019 May 3. PMID 31139321
- [Background] Zhang X, Rhoades J, Caan BJ, Cohn DE, Salani R, Noria S, Suarez AA, Paskett ED, Felix AS. Intentional weight loss, weight cycling, and endometrial cancer risk: a systematic review and meta-analysis. Int J Gynecol Cancer. 2019 Nov;29(9):1361-1371. doi: 10.1136/ijgc-2019-000728. Epub 2019 Aug 26. PMID 31451560
- [Background] Boyd P, O'Connor SG, Heckman-Stoddard BM, Sauter ER. Time-Restricted Feeding Studies and Possible Human Benefit. JNCI Cancer Spectr. 2022 May 2;6(3):pkac032. doi: 10.1093/jncics/pkac032. PMID 35657339
- [Background] Patterson RE, Sears DD. Metabolic Effects of Intermittent Fasting. Annu Rev Nutr. 2017 Aug 21;37:371-393. doi: 10.1146/annurev-nutr-071816-064634. Epub 2017 Jul 17. PMID 28715993
- [Background] Lee SA, Sypniewski C, Bensadon BA, McLaren C, Donahoo WT, Sibille KT, Anton S. Determinants of Adherence in Time-Restricted Feeding in Older Adults: Lessons from a Pilot Study. Nutrients. 2020 Mar 24;12(3):874. doi: 10.3390/nu12030874. PMID 32213965
- [Background] Anton SD, Lee SA, Donahoo WT, McLaren C, Manini T, Leeuwenburgh C, Pahor M. The Effects of Time Restricted Feeding on Overweight, Older Adults: A Pilot Study. Nutrients. 2019 Jun 30;11(7):1500. doi: 10.3390/nu11071500. PMID 31262054
- [Background] Gill S, Panda S. A Smartphone App Reveals Erratic Diurnal Eating Patterns in Humans that Can Be Modulated for Health Benefits. Cell Metab. 2015 Nov 3;22(5):789-98. doi: 10.1016/j.cmet.2015.09.005. Epub 2015 Sep 24. PMID 26411343
- [Background] Kahleova H, Lloren JI, Mashchak A, Hill M, Fraser GE. Meal Frequency and Timing Are Associated with Changes in Body Mass Index in Adventist Health Study 2. J Nutr. 2017 Sep;147(9):1722-1728. doi: 10.3945/jn.116.244749. Epub 2017 Jul 12. PMID 28701389
- [Background] Manoogian ENC, Panda S. Circadian rhythms, time-restricted feeding, and healthy aging. Ageing Res Rev. 2017 Oct;39:59-67. doi: 10.1016/j.arr.2016.12.006. Epub 2016 Dec 23. PMID 28017879
- [Background] Marinac CR, Natarajan L, Sears DD, Gallo LC, Hartman SJ, Arredondo E, Patterson RE. Prolonged Nightly Fasting and Breast Cancer Risk: Findings from NHANES (2009-2010). Cancer Epidemiol Biomarkers Prev. 2015 May;24(5):783-9. doi: 10.1158/1055-9965.EPI-14-1292. Epub 2015 Apr 20. PMID 25896523
- [Background] Zarrinpar A, Chaix A, Panda S. Daily Eating Patterns and Their Impact on Health and Disease. Trends Endocrinol Metab. 2016 Feb;27(2):69-83. doi: 10.1016/j.tem.2015.11.007. Epub 2015 Dec 17. PMID 26706567
- [Background] Di Francesco A, Di Germanio C, Bernier M, de Cabo R. A time to fast. Science. 2018 Nov 16;362(6416):770-775. doi: 10.1126/science.aau2095. PMID 30442801
- [Background] Shafi AA, Knudsen KE. Cancer and the Circadian Clock. Cancer Res. 2019 Aug 1;79(15):3806-3814. doi: 10.1158/0008-5472.CAN-19-0566. Epub 2019 Jul 12. PMID 31300477
- [Background] Jamshed H, Beyl RA, Della Manna DL, Yang ES, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves 24-Hour Glucose Levels and Affects Markers of the Circadian Clock, Aging, and Autophagy in Humans. Nutrients. 2019 May 30;11(6):1234. doi: 10.3390/nu11061234. PMID 31151228
- [Background] Wehrens SMT, Christou S, Isherwood C, Middleton B, Gibbs MA, Archer SN, Skene DJ, Johnston JD. Meal Timing Regulates the Human Circadian System. Curr Biol. 2017 Jun 19;27(12):1768-1775.e3. doi: 10.1016/j.cub.2017.04.059. Epub 2017 Jun 1. PMID 28578930
- [Background] Chaix A, Lin T, Le HD, Chang MW, Panda S. Time-Restricted Feeding Prevents Obesity and Metabolic Syndrome in Mice Lacking a Circadian Clock. Cell Metab. 2019 Feb 5;29(2):303-319.e4. doi: 10.1016/j.cmet.2018.08.004. Epub 2018 Aug 30. PMID 30174302
- [Background] Chaix A, Zarrinpar A, Miu P, Panda S. Time-restricted feeding is a preventative and therapeutic intervention against diverse nutritional challenges. Cell Metab. 2014 Dec 2;20(6):991-1005. doi: 10.1016/j.cmet.2014.11.001. PMID 25470547
- [Background] Gabel K, Hoddy KK, Haggerty N, Song J, Kroeger CM, Trepanowski JF, Panda S, Varady KA. Effects of 8-hour time restricted feeding on body weight and metabolic disease risk factors in obese adults: A pilot study. Nutr Healthy Aging. 2018 Jun 15;4(4):345-353. doi: 10.3233/NHA-170036. PMID 29951594
- [Background] Antonini A, Gentile G, Giglio M, Marcante A, Gage H, Touray MML, Fotiadis DI, Gatsios D, Konitsiotis S, Timotijevic L, Egan B, Hodgkins C, Biundo R, Pellicano C; PD_Manager consortium. Acceptability to patients, carers and clinicians of an mHealth platform for the management of Parkinson's disease (PD_Manager): study protocol for a pilot randomised controlled trial. Trials. 2018 Sep 14;19(1):492. doi: 10.1186/s13063-018-2767-4. PMID 30217235
- [Background] Arnason TG, Bowen MW, Mansell KD. Effects of intermittent fasting on health markers in those with type 2 diabetes: A pilot study. World J Diabetes. 2017 Apr 15;8(4):154-164. doi: 10.4239/wjd.v8.i4.154. PMID 28465792
- [Background] Kesztyus D, Cermak P, Gulich M, Kesztyus T. Adherence to Time-Restricted Feeding and Impact on Abdominal Obesity in Primary Care Patients: Results of a Pilot Study in a Pre-Post Design. Nutrients. 2019 Nov 21;11(12):2854. doi: 10.3390/nu11122854. PMID 31766465
- [Background] Marinac CR, Nelson SH, Breen CI, Hartman SJ, Natarajan L, Pierce JP, Flatt SW, Sears DD, Patterson RE. Prolonged Nightly Fasting and Breast Cancer Prognosis. JAMA Oncol. 2016 Aug 1;2(8):1049-55. doi: 10.1001/jamaoncol.2016.0164. PMID 27032109
- [Background] McAllister MJ, Pigg BL, Renteria LI, Waldman HS. Time-restricted feeding improves markers of cardiometabolic health in physically active college-age men: a 4-week randomized pre-post pilot study. Nutr Res. 2020 Mar;75:32-43. doi: 10.1016/j.nutres.2019.12.001. Epub 2019 Dec 4. PMID 31955013
- [Background] Carlson O, Martin B, Stote KS, Golden E, Maudsley S, Najjar SS, Ferrucci L, Ingram DK, Longo DL, Rumpler WV, Baer DJ, Egan J, Mattson MP. Impact of reduced meal frequency without caloric restriction on glucose regulation in healthy, normal-weight middle-aged men and women. Metabolism. 2007 Dec;56(12):1729-34. doi: 10.1016/j.metabol.2007.07.018. PMID 17998028
- [Background] Tinsley GM, La Bounty PM. Effects of intermittent fasting on body composition and clinical health markers in humans. Nutr Rev. 2015 Oct;73(10):661-74. doi: 10.1093/nutrit/nuv041. Epub 2015 Sep 15. PMID 26374764
- [Background] Wilkinson MJ, Manoogian ENC, Zadourian A, Lo H, Fakhouri S, Shoghi A, Wang X, Fleischer JG, Navlakha S, Panda S, Taub PR. Ten-Hour Time-Restricted Eating Reduces Weight, Blood Pressure, and Atherogenic Lipids in Patients with Metabolic Syndrome. Cell Metab. 2020 Jan 7;31(1):92-104.e5. doi: 10.1016/j.cmet.2019.11.004. Epub 2019 Dec 5. PMID 31813824
- [Background] Melkani GC, Panda S. Time-restricted feeding for prevention and treatment of cardiometabolic disorders. J Physiol. 2017 Jun 15;595(12):3691-3700. doi: 10.1113/JP273094. Epub 2017 Apr 25. PMID 28295377
- [Background] Hatori M, Vollmers C, Zarrinpar A, DiTacchio L, Bushong EA, Gill S, Leblanc M, Chaix A, Joens M, Fitzpatrick JA, Ellisman MH, Panda S. Time-restricted feeding without reducing caloric intake prevents metabolic diseases in mice fed a high-fat diet. Cell Metab. 2012 Jun 6;15(6):848-60. doi: 10.1016/j.cmet.2012.04.019. Epub 2012 May 17. PMID 22608008
- [Background] Mattson MP, Allison DB, Fontana L, Harvie M, Longo VD, Malaisse WJ, Mosley M, Notterpek L, Ravussin E, Scheer FA, Seyfried TN, Varady KA, Panda S. Meal frequency and timing in health and disease. Proc Natl Acad Sci U S A. 2014 Nov 25;111(47):16647-53. doi: 10.1073/pnas.1413965111. Epub 2014 Nov 17. PMID 25404320
- [Background] Sundaram S, Yan L. Time-restricted feeding mitigates high-fat diet-enhanced mammary tumorigenesis in MMTV-PyMT mice. Nutr Res. 2018 Nov;59:72-79. doi: 10.1016/j.nutres.2018.07.014. Epub 2018 Jul 31. PMID 30442235
- [Background] Gabel K, Hoddy KK, Varady KA. Safety of 8-h time restricted feeding in adults with obesity. Appl Physiol Nutr Metab. 2019 Jan;44(1):107-109. doi: 10.1139/apnm-2018-0389. Epub 2018 Sep 14. PMID 30216730
- [Background] Sutton EF, Beyl R, Early KS, Cefalu WT, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves Insulin Sensitivity, Blood Pressure, and Oxidative Stress Even without Weight Loss in Men with Prediabetes. Cell Metab. 2018 Jun 5;27(6):1212-1221.e3. doi: 10.1016/j.cmet.2018.04.010. Epub 2018 May 10. PMID 29754952
- [Background] Harvie MN, Pegington M, Mattson MP, Frystyk J, Dillon B, Evans G, Cuzick J, Jebb SA, Martin B, Cutler RG, Son TG, Maudsley S, Carlson OD, Egan JM, Flyvbjerg A, Howell A. The effects of intermittent or continuous energy restriction on weight loss and metabolic disease risk markers: a randomized trial in young overweight women. Int J Obes (Lond). 2011 May;35(5):714-27. doi: 10.1038/ijo.2010.171. Epub 2010 Oct 5. PMID 20921964
- [Background] Gasmi M, Sellami M, Denham J, Padulo J, Kuvacic G, Selmi W, Khalifa R. Time-restricted feeding influences immune responses without compromising muscle performance in older men. Nutrition. 2018 Jul-Aug;51-52:29-37. doi: 10.1016/j.nut.2017.12.014. Epub 2018 Feb 3. PMID 29571007
- [Background] Moro T, Tinsley G, Bianco A, Marcolin G, Pacelli QF, Battaglia G, Palma A, Gentil P, Neri M, Paoli A. Effects of eight weeks of time-restricted feeding (16/8) on basal metabolism, maximal strength, body composition, inflammation, and cardiovascular risk factors in resistance-trained males. J Transl Med. 2016 Oct 13;14(1):290. doi: 10.1186/s12967-016-1044-0. PMID 27737674
- [Background] Ravussin E, Beyl RA, Poggiogalle E, Hsia DS, Peterson CM. Early Time-Restricted Feeding Reduces Appetite and Increases Fat Oxidation But Does Not Affect Energy Expenditure in Humans. Obesity (Silver Spring). 2019 Aug;27(8):1244-1254. doi: 10.1002/oby.22518. PMID 31339000
- [Background] Lowe DA, Wu N, Rohdin-Bibby L, Moore AH, Kelly N, Liu YE, Philip E, Vittinghoff E, Heymsfield SB, Olgin JE, Shepherd JA, Weiss EJ. Effects of Time-Restricted Eating on Weight Loss and Other Metabolic Parameters in Women and Men With Overweight and Obesity: The TREAT Randomized Clinical Trial. JAMA Intern Med. 2020 Nov 1;180(11):1491-1499. doi: 10.1001/jamainternmed.2020.4153. PMID 32986097
- [Background] Hutchison AT, Liu B, Wood RE, Vincent AD, Thompson CH, O'Callaghan NJ, Wittert GA, Heilbronn LK. Effects of Intermittent Versus Continuous Energy Intakes on Insulin Sensitivity and Metabolic Risk in Women with Overweight. Obesity (Silver Spring). 2019 Jan;27(1):50-58. doi: 10.1002/oby.22345. PMID 30569640
- [Background] Parr EB, Devlin BL, Radford BE, Hawley JA. A Delayed Morning and Earlier Evening Time-Restricted Feeding Protocol for Improving Glycemic Control and Dietary Adherence in Men with Overweight/Obesity: A Randomized Controlled Trial. Nutrients. 2020 Feb 17;12(2):505. doi: 10.3390/nu12020505. PMID 32079327
- [Background] Adafer R, Messaadi W, Meddahi M, Patey A, Haderbache A, Bayen S, Messaadi N. Food Timing, Circadian Rhythm and Chrononutrition: A Systematic Review of Time-Restricted Eating's Effects on Human Health. Nutrients. 2020 Dec 8;12(12):3770. doi: 10.3390/nu12123770. PMID 33302500
- [Background] He M, Wang J, Liang Q, Li M, Guo H, Wang Y, Deji C, Sui J, Wang YW, Liu Y, Zheng Y, Qian B, Chen H, Ma M, Su S, Geng H, Zhou WX, Guo X, Zhu WZ, Zhang M, Chen Z, Rensen PCN, Hui CC, Wang Y, Shi B. Time-restricted eating with or without low-carbohydrate diet reduces visceral fat and improves metabolic syndrome: A randomized trial. Cell Rep Med. 2022 Oct 18;3(10):100777. doi: 10.1016/j.xcrm.2022.100777. Epub 2022 Oct 10. PMID 36220069
- [Background] Thomas EA, Zaman A, Sloggett KJ, Steinke S, Grau L, Catenacci VA, Cornier MA, Rynders CA. Early time-restricted eating compared with daily caloric restriction: A randomized trial in adults with obesity. Obesity (Silver Spring). 2022 May;30(5):1027-1038. doi: 10.1002/oby.23420. PMID 35470974
- [Background] Lin S, Cienfuegos S, Ezpeleta M, Gabel K, Pavlou V, Mulas A, Chakos K, McStay M, Wu J, Tussing-Humphreys L, Alexandria SJ, Sanchez J, Unterman T, Varady KA. Time-Restricted Eating Without Calorie Counting for Weight Loss in a Racially Diverse Population : A Randomized Controlled Trial. Ann Intern Med. 2023 Jul;176(7):885-895. doi: 10.7326/M23-0052. Epub 2023 Jun 27. PMID 37364268
- [Background] Faris MA, Kacimi S, Al-Kurd RA, Fararjeh MA, Bustanji YK, Mohammad MK, Salem ML. Intermittent fasting during Ramadan attenuates proinflammatory cytokines and immune cells in healthy subjects. Nutr Res. 2012 Dec;32(12):947-55. doi: 10.1016/j.nutres.2012.06.021. Epub 2012 Oct 4. PMID 23244540
- [Background] Almeneessier AS, BaHammam AA, Alzoghaibi M, Olaish AH, Nashwan SZ, BaHammam AS. The effects of diurnal intermittent fasting on proinflammatory cytokine levels while controlling for sleep/wake pattern, meal composition and energy expenditure. PLoS One. 2019 Dec 10;14(12):e0226034. doi: 10.1371/journal.pone.0226034. eCollection 2019. PMID 31821377
- [Background] Mindikoglu AL, Park J, Opekun AR, Abdulsada MM, Wilhelm ZR, Jalal PK, Devaraj S, Jung SY. Dawn-to-dusk dry fasting induces anti-atherosclerotic, anti-inflammatory, and anti-tumorigenic proteome in peripheral blood mononuclear cells in subjects with metabolic syndrome. Metabol Open. 2022 Nov 1;16:100214. doi: 10.1016/j.metop.2022.100214. eCollection 2022 Dec. PMID 36506940
- [Background] Marinac CR, Sears DD, Natarajan L, Gallo LC, Breen CI, Patterson RE. Frequency and Circadian Timing of Eating May Influence Biomarkers of Inflammation and Insulin Resistance Associated with Breast Cancer Risk. PLoS One. 2015 Aug 25;10(8):e0136240. doi: 10.1371/journal.pone.0136240. eCollection 2015. PMID 26305095
- [Background] Wirth MD, Zhao L, Turner-McGrievy GM, Ortaglia A. Associations between Fasting Duration, Timing of First and Last Meal, and Cardiometabolic Endpoints in the National Health and Nutrition Examination Survey. Nutrients. 2021 Aug 3;13(8):2686. doi: 10.3390/nu13082686. PMID 34444846
- [Background] Das M, Webster NJG. Obesity, cancer risk, and time-restricted eating. Cancer Metastasis Rev. 2022 Sep;41(3):697-717. doi: 10.1007/s10555-022-10061-3. Epub 2022 Aug 19. PMID 35984550
- [Background] Guinter MA, Campbell PT, Patel AV, McCullough ML. Irregularity in breakfast consumption and daily meal timing patterns in association with body weight status and inflammation. Br J Nutr. 2019 Nov 28;122(10):1192-1200. doi: 10.1017/S0007114519002125. Epub 2019 Aug 20. PMID 31637978
- [Background] Srour B P-CA, Fezeu LK, Julia C, Bellicha A, Kesse-Guyot E, Romaguera D, Kogevinas M, Touvier M. Circadian nutritional behaviours and risk of type 2 diabetes in NutriNet-Santé. Eur J Clin Nutr. 2022;32(Supplement 3).
- [Background] Pearson-Stuttard J, Papadimitriou N, Markozannes G, Cividini S, Kakourou A, Gill D, Rizos EC, Monori G, Ward HA, Kyrgiou M, Gunter MJ, Tsilidis KK. Type 2 Diabetes and Cancer: An Umbrella Review of Observational and Mendelian Randomization Studies. Cancer Epidemiol Biomarkers Prev. 2021 Jun;30(6):1218-1228. doi: 10.1158/1055-9965.EPI-20-1245. Epub 2021 Mar 18. PMID 33737302
- [Background] Srour B, Plancoulaine S, Andreeva VA, Fassier P, Julia C, Galan P, Hercberg S, Deschasaux M, Latino-Martel P, Touvier M. Circadian nutritional behaviours and cancer risk: New insights from the NutriNet-sante prospective cohort study: Disclaimers. Int J Cancer. 2018 Nov 15;143(10):2369-2379. doi: 10.1002/ijc.31584. Epub 2018 Jul 3. PMID 29744870
- [Background] Kogevinas M, Espinosa A, Castello A, Gomez-Acebo I, Guevara M, Martin V, Amiano P, Alguacil J, Peiro R, Moreno V, Costas L, Fernandez-Tardon G, Jimenez JJ, Marcos-Gragera R, Perez-Gomez B, Llorca J, Moreno-Iribas C, Fernandez-Villa T, Oribe M, Aragones N, Papantoniou K, Pollan M, Castano-Vinyals G, Romaguera D. Effect of mistimed eating patterns on breast and prostate cancer risk (MCC-Spain Study). Int J Cancer. 2018 Nov 15;143(10):2380-2389. doi: 10.1002/ijc.31649. Epub 2018 Jul 17. PMID 30016830
- [Background] Palomar-Cros A, Espinosa A, Straif K, Perez-Gomez B, Papantoniou K, Gomez-Acebo I, Molina-Barcelo A, Olmedo-Requena R, Alguacil J, Fernandez-Tardon G, Casabonne D, Aragones N, Castano-Vinyals G, Pollan M, Romaguera D, Kogevinas M. The Association of Nighttime Fasting Duration and Prostate Cancer Risk: Results from the Multicase-Control (MCC) Study in Spain. Nutrients. 2021 Jul 30;13(8):2662. doi: 10.3390/nu13082662. PMID 34444822
- [Background] Long CR, Rowland B, McElfish PA, Ayers BL, Narcisse MR. Food Security Status of Native Hawaiians and Pacific Islanders in the US: Analysis of a National Survey. J Nutr Educ Behav. 2020 Aug;52(8):788-795. doi: 10.1016/j.jneb.2020.01.009. Epub 2020 Mar 14. PMID 32184077
- [Background] Rabaut LJ. Medically Tailored Meals as a Prescription for Treatment of Food-Insecure Type 2 Diabetics. J Patient Cent Res Rev. 2019 Apr 29;6(2):179-183. doi: 10.17294/2330-0698.1693. eCollection 2019 Spring. PMID 31414029
- [Background] Berkowitz SA, Terranova J, Randall L, Cranston K, Waters DB, Hsu J. Association Between Receipt of a Medically Tailored Meal Program and Health Care Use. JAMA Intern Med. 2019 Jun 1;179(6):786-793. doi: 10.1001/jamainternmed.2019.0198. PMID 31009050
- [Background] Berkowitz SA, Delahanty LM, Terranova J, Steiner B, Ruazol MP, Singh R, Shahid NN, Wexler DJ. Medically Tailored Meal Delivery for Diabetes Patients with Food Insecurity: a Randomized Cross-over Trial. J Gen Intern Med. 2019 Mar;34(3):396-404. doi: 10.1007/s11606-018-4716-z. Epub 2018 Nov 12. PMID 30421335
- [Background] Hager K, Cudhea FP, Wong JB, Berkowitz SA, Downer S, Lauren BN, Mozaffarian D. Association of National Expansion of Insurance Coverage of Medically Tailored Meals With Estimated Hospitalizations and Health Care Expenditures in the US. JAMA Netw Open. 2022 Oct 3;5(10):e2236898. doi: 10.1001/jamanetworkopen.2022.36898. PMID 36251292
- [Background] McElfish PA, Long CR, Kaholokula JK, Aitaoto N, Bursac Z, Capelle L, Laelan M, Bing WI, Riklon S, Rowland B, Ayers BL, Wilmoth RO, Langston KN, Schootman M, Selig JP, Yeary KHK. Design of a comparative effectiveness randomized controlled trial testing a faith-based Diabetes Prevention Program (WORD DPP) vs. a Pacific culturally adapted Diabetes Prevention Program (PILI DPP) for Marshallese in the United States. Medicine (Baltimore). 2018 May;97(19):e0677. doi: 10.1097/MD.0000000000010677. PMID 29742712
- [Background] DePue JD, Rosen RK, Seiden A, Bereolos N, Chima ML, Goldstein MG, Nu'usolia O, Tuitele J, McGarvey ST. Implementation of a culturally tailored diabetes intervention with community health workers in American Samoa. Diabetes Educ. 2013 Nov-Dec;39(6):761-71. doi: 10.1177/0145721713504630. Epub 2013 Sep 19. PMID 24052204
- [Background] Palu E, MacMillan DF, McBride DKA, Thomson DR, Zarora R, Simmons D. Effects of lifestyle interventions on weight amongst Pasifika communities: A systematic review and meta-analysis. Lancet Reg Health West Pac. 2022 May 31;25:100483. doi: 10.1016/j.lanwpc.2022.100483. eCollection 2022 Aug. PMID 35669931
- [Background] Kaholokula JK, Kekauoha P, Dillard A, Yoshimura S, Palakiko DM, Hughes C, Townsend CK. The PILI 'Ohana Project: a community-academic partnership to achieve metabolic health equity in Hawai'i. Hawaii J Med Public Health. 2014 Dec;73(12 Suppl 3):29-33. PMID 25535599
- [Background] Kaholokula JK, Mau MK, Efird JT, Leake A, West M, Palakiko DM, Yoshimura SR, Kekauoha BP, Rose C, Gomes H. A family and community focused lifestyle program prevents weight regain in Pacific Islanders: a pilot randomized controlled trial. Health Educ Behav. 2012 Aug;39(4):386-95. doi: 10.1177/1090198110394174. Epub 2011 May 6. PMID 21551421
- [Background] Phillips NE, Mareschal J, Schwab N, Manoogian ENC, Borloz S, Ostinelli G, Gauthier-Jaques A, Umwali S, Gonzalez Rodriguez E, Aeberli D, Hans D, Panda S, Rodondi N, Naef F, Collet TH. The Effects of Time-Restricted Eating versus Standard Dietary Advice on Weight, Metabolic Health and the Consumption of Processed Food: A Pragmatic Randomised Controlled Trial in Community-Based Adults. Nutrients. 2021 Mar 23;13(3):1042. doi: 10.3390/nu13031042. PMID 33807102
- [Background] Xiao Q, Bauer C, Layne T, Playdon M. The association between overnight fasting and body mass index in older adults: the interaction between duration and timing. Int J Obes (Lond). 2021 Mar;45(3):555-564. doi: 10.1038/s41366-020-00715-z. Epub 2020 Nov 19. PMID 33214704
- [Background] Schatzkin A, Subar AF, Thompson FE, Harlan LC, Tangrea J, Hollenbeck AR, Hurwitz PE, Coyle L, Schussler N, Michaud DS, Freedman LS, Brown CC, Midthune D, Kipnis V. Design and serendipity in establishing a large cohort with wide dietary intake distributions : the National Institutes of Health-American Association of Retired Persons Diet and Health Study. Am J Epidemiol. 2001 Dec 15;154(12):1119-25. doi: 10.1093/aje/154.12.1119. PMID 11744517
- [Background] US Department of Health and Human Services Office of Minority Health. Profile: Native Hawaiians/Pacific Islanders 2019 [Accessed 9th October, 2019]. Available from: https://minorityhealth.hhs.gov/omh/browse.aspx?lvl=3&lvlid=65
- [Background] HJ A. Doing qualitative research in education settings. . Albany: State University of New York Press; 2002.
- [Background] Roenneberg T, Keller LK, Fischer D, Matera JL, Vetter C, Winnebeck EC. Human activity and rest in situ. Methods Enzymol. 2015;552:257-83. doi: 10.1016/bs.mie.2014.11.028. Epub 2015 Jan 5. PMID 25707281
- [Background] Matthews CE, Keadle SK, Sampson J, Lyden K, Bowles HR, Moore SC, Libertine A, Freedson PS, Fowke JH. Validation of a previous-day recall measure of active and sedentary behaviors. Med Sci Sports Exerc. 2013 Aug;45(8):1629-38. doi: 10.1249/MSS.0b013e3182897690. PMID 23863547
- [Background] Fleischer JG, Das SK, Bhapkar M, Manoogian ENC, Panda S. Associations between the timing of eating and weight-loss in calorically restricted healthy adults: Findings from the CALERIE study. Exp Gerontol. 2022 Aug;165:111837. doi: 10.1016/j.exger.2022.111837. Epub 2022 May 20. PMID 35598698
- [Background] Dossus L, Kouloura E, Biessy C, Viallon V, Siskos AP, Dimou N, Rinaldi S, Merritt MA, Allen N, Fortner R, Kaaks R, Weiderpass E, Gram IT, Rothwell JA, Lecuyer L, Severi G, Schulze MB, Nost TH, Crous-Bou M, Sanchez MJ, Amiano P, Colorado-Yohar SM, Gurrea AB, Schmidt JA, Palli D, Agnoli C, Tumino R, Sacerdote C, Mattiello A, Vermeulen R, Heath AK, Christakoudi S, Tsilidis KK, Travis RC, Gunter MJ, Keun HC. Prospective analysis of circulating metabolites and endometrial cancer risk. Gynecol Oncol. 2021 Aug;162(2):475-481. doi: 10.1016/j.ygyno.2021.06.001. Epub 2021 Jun 5. PMID 34099314
- [Background] Moore SC, Mazzilli KM, Sampson JN, Matthews CE, Carter BD, Playdon MC, Wang Y, Stevens VL. A Metabolomics Analysis of Postmenopausal Breast Cancer Risk in the Cancer Prevention Study II. Metabolites. 2021 Feb 10;11(2):95. doi: 10.3390/metabo11020095. PMID 33578791
- [Background] Moore SC, Playdon MC, Sampson JN, Hoover RN, Trabert B, Matthews CE, Ziegler RG. A Metabolomics Analysis of Body Mass Index and Postmenopausal Breast Cancer Risk. J Natl Cancer Inst. 2018 Jun 1;110(6):588-597. doi: 10.1093/jnci/djx244. PMID 29325144
- [Background] Playdon MC, Ziegler RG, Sampson JN, Stolzenberg-Solomon R, Thompson HJ, Irwin ML, Mayne ST, Hoover RN, Moore SC. Nutritional metabolomics and breast cancer risk in a prospective study. Am J Clin Nutr. 2017 Aug;106(2):637-649. doi: 10.3945/ajcn.116.150912. Epub 2017 Jun 28. PMID 28659298
- [Background] Ruijgrok C, Dekker JM, Beulens JW, Brouwer IA, Coupe VMH, Heymans MW, Sijtsma FPC, Mela DJ, Zock PL, Olthof MR, Alssema M. Size and shape of the associations of glucose, HbA1c, insulin and HOMA-IR with incident type 2 diabetes: the Hoorn Study. Diabetologia. 2018 Jan;61(1):93-100. doi: 10.1007/s00125-017-4452-7. Epub 2017 Oct 10. PMID 29018885
- [Background] Winn M, Karra P, Freisling H, Gunter MJ, Haaland B, Litchman ML, Doherty JA, Playdon MC, Hardikar S. Metabolic obesity phenotypes and obesity-related cancer risk in the National Health and Nutrition Examination Survey. Endocrinol Diabetes Metab. 2023 Jul;6(4):e433. doi: 10.1002/edm2.433. Epub 2023 Jun 5. PMID 37277888
- [Background] Inc. LS. LabVantage 2023 [Accessed September 10th, 2023]. Available from: https://www.labvantage.com/.
- [Background] Kaholokula JK, Wilson RE, Townsend CK, Zhang GX, Chen J, Yoshimura SR, Dillard A, Yokota JW, Palakiko DM, Gamiao S, Hughes CK, Kekauoha BK, Mau MK. Translating the Diabetes Prevention Program in Native Hawaiian and Pacific Islander communities: the PILI 'Ohana Project. Transl Behav Med. 2014 Jun;4(2):149-59. doi: 10.1007/s13142-013-0244-x. PMID 24904698
- [Background] Baranowski T PC, Parcel, GS. Health Behavior and Health Education: Theory, Research, and Practice. San Francisco Jossey-Bass; 2003.
- [Background] Matenga-Ikihele A, McCool J, Dobson R, Fa'alau F, Whittaker R. The characteristics of behaviour change interventions used among Pacific people: a systematic search and narrative synthesis. BMC Public Health. 2021 Mar 4;21(1):435. doi: 10.1186/s12889-021-10420-9. PMID 33663438
- [Background] Yang KI, Chung-Do JJ, Fujitani L, Foster A, Mark S, Okada Y, Saad-Jube Z, Youkhana F, Braun KL, Cassel K, Helm S, Ka'opua LS, Mataira PJ, Nishita C, Okamoto SK, Ing CT, Qureshi K, Umemoto K. Advancing Community-Based Participatory Research to Address Health Disparities in Hawai'i: Perspectives from Academic Researchers. Hawaii J Med Public Health. 2019 Mar;78(3):83-88. PMID 30854253
- [Background] Campbell PT, Newton CC, Jacobs EJ, McCullough ML, Wang Y, Rees-Punia E, Guinter MA, Murphy N, Koshiol J, Dehal AN, Rohan T, Strickler H, Petrick J, Gunter M, Zhang X, McGlynn KA, Pollak M, Patel AV, Gapstur SM. Prospective associations of hemoglobin A1c and c-peptide with risk of diabetes-related cancers in the Cancer Prevention Study-II Nutrition Cohort. Cancer Res Commun. 2022 Jul;2(7):653-662. doi: 10.1158/2767-9764.crc-22-0082. Epub 2022 Jul 14. PMID 36712480
- [Background] Murphy N, Cross AJ, Abubakar M, Jenab M, Aleksandrova K, Boutron-Ruault MC, Dossus L, Racine A, Kuhn T, Katzke VA, Tjonneland A, Petersen KE, Overvad K, Quiros JR, Jakszyn P, Molina-Montes E, Dorronsoro M, Huerta JM, Barricarte A, Khaw KT, Wareham N, Travis RC, Trichopoulou A, Lagiou P, Trichopoulos D, Masala G, Krogh V, Tumino R, Vineis P, Panico S, Bueno-de-Mesquita HB, Siersema PD, Peeters PH, Ohlsson B, Ericson U, Palmqvist R, Nystrom H, Weiderpass E, Skeie G, Freisling H, Kong SY, Tsilidis K, Muller DC, Riboli E, Gunter MJ. A Nested Case-Control Study of Metabolically Defined Body Size Phenotypes and Risk of Colorectal Cancer in the European Prospective Investigation into Cancer and Nutrition (EPIC). PLoS Med. 2016 Apr 5;13(4):e1001988. doi: 10.1371/journal.pmed.1001988. eCollection 2016 Apr. PMID 27046222
- [Background] ARUP. ARUP Laboratories 2023 [Accessed September 9th, 2023]. Available from: https://www.aruplab.com/
- [Background] Xia J, Wishart DS. Using MetaboAnalyst 3.0 for Comprehensive Metabolomics Data Analysis. Curr Protoc Bioinformatics. 2016 Sep 7;55:14.10.1-14.10.91. doi: 10.1002/cpbi.11. PMID 27603023
- [Background] Kirwan JA, Brennan L, Broadhurst D, Fiehn O, Cascante M, Dunn WB, Schmidt MA, Velagapudi V. Preanalytical Processing and Biobanking Procedures of Biological Samples for Metabolomics Research: A White Paper, Community Perspective (for "Precision Medicine and Pharmacometabolomics Task Group"-The Metabolomics Society Initiative). Clin Chem. 2018 Aug;64(8):1158-1182. doi: 10.1373/clinchem.2018.287045. Epub 2018 Jun 19. PMID 29921725
- [Background] MSI Board Members; Sansone SA, Fan T, Goodacre R, Griffin JL, Hardy NW, Kaddurah-Daouk R, Kristal BS, Lindon J, Mendes P, Morrison N, Nikolau B, Robertson D, Sumner LW, Taylor C, van der Werf M, van Ommen B, Fiehn O. The metabolomics standards initiative. Nat Biotechnol. 2007 Aug;25(8):846-8. doi: 10.1038/nbt0807-846b. No abstract available. PMID 17687353
- [Background] Zheng Y, Klem ML, Sereika SM, Danford CA, Ewing LJ, Burke LE. Self-weighing in weight management: a systematic literature review. Obesity (Silver Spring). 2015 Feb;23(2):256-65. doi: 10.1002/oby.20946. Epub 2014 Dec 17. PMID 25521523
- [Background] Robinson KA, Dinglas VD, Sukrithan V, Yalamanchilli R, Mendez-Tellez PA, Dennison-Himmelfarb C, Needham DM. Updated systematic review identifies substantial number of retention strategies: using more strategies retains more study participants. J Clin Epidemiol. 2015 Dec;68(12):1481-7. doi: 10.1016/j.jclinepi.2015.04.013. Epub 2015 Jun 10. PMID 26186981
- [Background] Abshire M, Dinglas VD, Cajita MI, Eakin MN, Needham DM, Himmelfarb CD. Participant retention practices in longitudinal clinical research studies with high retention rates. BMC Med Res Methodol. 2017 Feb 20;17(1):30. doi: 10.1186/s12874-017-0310-z. PMID 28219336
- [Background] Braun V, & Clarke, V. . Thematic analysis. In: H. Cooper MNC, L. M. McMullen, A. T. Panter, D. Rindskopf, & K. J. Sher (Eds.), editor. APA handbook of research methods in psychology: Research designs: Quantitative, qualitative, neuropsychological, and biological Washington, DC American Psychological Association; 2023.
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c332. doi: 10.1136/bmj.c332. PMID 20332509